CLINICAL TRIAL: NCT05141006
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled, Parallel Arm Study to Assess the Safety and Efficacy of a Single Treatment of BOTOX, Followed by an Optional Open-Label Treatment With BOTOX, in Female Subjects With Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS)
Brief Title: Study of BOTOX Injections to Assess Change in Disease Activity and Adverse Events in Adult Female Participants With Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS)
Acronym: IC/BPS POC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M21-459
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS)
Keywords: Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS); BOTOX; Botulinum Toxin Type A; OnabotulinumtoxinA
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BOTOX (Experimental): Participants will receive BOTOX on Day 1 and will be followed for at least 12 weeks in treatment period 1. An optional dose of BOTOX in Treatment 2 can be requested between Weeks 12 and 24.
  Interventions: Drug: BOTOX
- Placebo (Placebo Comparator): Participants will receive placebo on Day 1 and will be followed for at least 12 weeks in treatment period 1. An optional dose of BOTOX in Treatment 2 can be requested between Weeks 12 and 24.
  Interventions: Drug: BOTOX; Drug: Placebo for BOTOX

INTERVENTIONS:
Drug: BOTOX — Injection into the bladder
  Other Names: OnabotulinumtoxinA; Botulinum Toxin Type A
Drug: Placebo for BOTOX — Injection into the bladder
  Arms: Placebo

SUMMARY:
Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) is a chronic and debilitating urological complex of disorders characterized by symptoms of bladder pain or discomfort, mostly upon bladder filling, and often accompanied by lower urinary tract symptoms (LUTS). This study will assess how safe and effective BOTOX (onabotulinumtoxinA) is in treating IC/BPS. Adverse events and change in disease symptoms will be evaluated.

BOTOX (onabotulinumtoxinA) is an investigational drug being developed for the treatment of Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS). Study doctors randomly assign the participants to 1 of 2 groups, called treatment arms, to receive BOTOX or placebo. There is a 1 in 2 chance that participants will be assigned to placebo. Approximately 80 female participants, aged 18 to 75 years, with a diagnosis of IC/BPS will be enrolled in approximately 40 sites in the United States and Canada.

Participants will receive BOTOX or placebo injected into the bladder on Day 1 and will be followed for at least 12 weeks in treatment 1. Eligible participants may request additional dose of BOTOX between Weeks 12 and 24, and will be followed for 12 weeks in treatment period 2.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

- Presence of Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) symptoms for at least 6 months, diagnosed by the investigator as IC/BPS, and confirmed dominant bladder derived pain.

Exclusion Criteria:

- History or current diagnosis of Hunner Lesions.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Change in Average Daily Worst Bladder Pain | Baseline (Week 0) to Week 6
  Daily worst bladder pain will be assessed on the 11-point (0-10) numeric rating scale where 0 = no pain and 10 = the worst pain possible.

SECONDARY OUTCOMES:
Change in the Average Number of Micturition Episodes per 24-hour Period | Baseline (Week 0) to Week 6
  Micturition (whether participant was able to urinate) episodes will be collected on the 3-day bladder diary.
Change in the Average Number of Urgency Episodes per 24-hour Period | Baseline (Week 0) to Week 6
  Urgency episodes will be reported in the 3-day bladder diary.
Change in the Average Number of Nocturia Episodes per 24-hour Period | Baseline (Week 0) to Week 6
  Nocturia episodes will be reported in the 3-day bladder diary.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (43):
- United States (40):
  - Urology Centers of Alabama /ID# 243600, Homewood, Alabama
  - Urology Associates of Mobile, PA /ID# 255854, Mobile, Alabama
  - Alliance for Multispecialty Research (AMR) - Mobile /ID# 241002, Mobile, Alabama
  - Sun Kim Urology /ID# 257566, Buena Park, California
  - Cedars-Sinai Medical Center /ID# 245786, Los Angeles, California
  - University of California, Los Angeles /ID# 245131, Los Angeles, California
  - Tri Valley Urology Medical Group /ID# 254918, Murrieta, California
  - Inland Urology /ID# 255410, Pomona, California
  - UCSD Medical Center /ID# 244935, San Diego, California
  - Prestige Medical Group /ID# 257564, Santa Ana, California
  - Hartford Healthcare Group - Farmington /ID# 241037, Farmington, Connecticut
  - Medstar Health Research Institute /ID# 245371, Washington D.C., District of Columbia
  - Manatee Medical Research Institute /ID# 243859, Bradenton, Florida
  - Clinical Research Center FL /ID# 243961, Pompano Beach, Florida
  - Ochsner LSU Health Shreveport - Regional Urology. /ID# 241034, Shreveport, Louisiana
  - Bay State Clincial Trials, Inc /ID# 240848, Watertown, Massachusetts
  - Sheldon Freedman MD, ltd /ID# 241003, Las Vegas, Nevada
  - Western New York Urology Associates - Harlem Professional Park /ID# 241036, Cheektowaga, New York
  - North Shore University Hospital /ID# 242594, New Hyde Park, New York
  - NYU Langone Medical Center /ID# 241090, New York, New York
  - Columbia University Medical Center /ID# 241086, New York, New York
  - Columbia University Medical Center /ID# 241087, New York, New York
  - Crystal Run Healthcare - Warwick /ID# 241116, Warwick, New York
  - Cleveland Clinic Avon Hospital /ID# 247221, Avon, Ohio
  - The Christ Hospital /ID# 244800, Cincinnati, Ohio
  - Univ Hosp Cleveland /ID# 247228, Cleveland, Ohio
  - MetroHealth Medical Center /ID# 254812, Cleveland, Ohio
  - Wright State Physicians Obstetrics and Gynecology /ID# 241112, Oakwood, Ohio
  - The Institute for Female Pelvic Medicine and Reconstructive Surgery - Allentown /ID# 241012, Allentown, Pennsylvania
  - MidLantic Urology /ID# 240997, Bala-Cynwyd, Pennsylvania
  - Thomas Jefferson University Hospital /ID# 243703, Philadelphia, Pennsylvania
  - Medical University of South Carolina /ID# 242780, Charleston, South Carolina
  - Southern Shores Urogynecology /ID# 253316, Myrtle Beach, South Carolina
  - Chattanooga Research and Medicine /ID# 241092, Chattanooga, Tennessee
  - Urology Associates PC - Nashville /ID# 242914, Nashville, Tennessee
  - University of Texas Southwestern Medical Center /ID# 244931, Dallas, Texas
  - Advances in Health, Inc. /ID# 240850, Pearland, Texas
  - Potomac Urology - Alexandria /ID# 243963, Alexandria, Virginia
  - Specialists For Women - Hillpoint /ID# 242541, Suffolk, Virginia
  - Urology of Virginia /ID# 240843, Virginia Beach, Virginia
- Canada (3):
  - Queen's University /ID# 243972, Kingston, Ontario
  - Sunnybrook Health Sciences Ctr /ID# 243243, Toronto, Ontario
  - CHUS - Hopital Fleurimont /ID# 244058, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/